CLINICAL TRIAL: NCT05622357
Title: Prospective Phase II Study of Hypofractionated Short Course Radiation Therapy Followed by Neoadjuvant Chemotherapy and Surgery in Locally Advanced Rectal Cancer
Brief Title: Prospective Study of Short Course Radiation Therapy Followed by Neoadjuvant Chemotherapy and Surgery in Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Yasser Anwar, Lecturer of Radiation Oncology, National Cancer Institute, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201617097
Record Dates: First submitted 2022-11-11; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Locally Advanced Rectal Carcinoma
Keywords: advanced rectal cancer- short course radiation - chemotherapy-surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short course RT followed by full course of chemotherapy then surgery (Experimental): Short course radiation therapy ( 25 Gy/ 5 fractions/ 1 week) , followed by 6 cycles of chemotherapy CAPOX, followed 4-6 weeks by surgery.
  Interventions: Radiation: short course radiation therapy followed by 6 cycles of CAPOX then surgery

INTERVENTIONS:
Radiation: short course radiation therapy followed by 6 cycles of CAPOX then surgery — Short course RT 5 x5 Gy followed by 6 cycles CAPOX then surgery

SUMMARY:
The goal of this clinical trial is to investigate total neoadjuvant therapy (TNT) using short course radiation therapy (SCRT) followed by full course of chemotherapy then surgery in locally advanced rectal cancer. The main questions it aims to answer are:

* Is total neoadjuvant treatment in this design safe & tolerable?
* Impact of this design on treatment related outcomes in terms of pathological and clinical responses.

DETAILED DESCRIPTION:
Patients will be assigned to an experimental arm in which preoperative short course 5 x 5 Gy radiation therapy is followed by six cycles of combination chemotherapy (capecitabine and oxaliplatin) and surgery within 4-6 weeks

ELIGIBILITY:
Inclusion Criteria:

* Histopathological proof of rectal adenocarcinoma.
* Tumors located within 15 cm and not less than 4 cm from anal verge.
* Age: ≥ 18 years.
* Locally advanced resectable rectal cancer (cT3/4 N0- Any T N+ve).
* ECOG Performance Status: 0-2.

Exclusion Criteria:

* Non-epithelial rectal malignancy such as sarcoma or lymphoma.
* Unresectable tumors in which surgery will never be possible even if substantial tumor downsizing is seen.
* Recurrent rectal cancer.
* Previous history of malignancy within the last 5 years.
* Previous pelvic irradiation.
* Psychiatric or addictive disorder that would preclude study therapy.
* Concurrent uncontrolled medical conditions.
* Pregnancy or breast feeding.
* Any contraindication to surgery.
* Extensive peripheral neuropathy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-03-18 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
pathological complete response (pCR) | within 30 days
  No residual disease in surgical specimen
clinical complete response(cCR) | within 30 days
  No residual disease after end of radiation and chemotherapy by examination,imaging and colonoscopy
Sphincter saving surgery | within 6 months
  Patients who were deemed abdomino-perineal resection before treatment start & were able to undergo low anterior resection after end of treatment

SECONDARY OUTCOMES:
Local control | 3 years
  defined as the period calculated from the date of end of treatment to the date of occurrence of loco-regional failure.
Overall survival | 3 years
  defined as period from diagnosis till last follow up or death from any cause
Disease free survival | within 3 years
  defined as the period calculated from the date of end of treatment to the date of occurrence of loco-regional failure or distant failure, whichever comes first.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Cairo, الجيزة, Egypt